CLINICAL TRIAL: NCT01412008
Title: Exploring Advanced Imaging Techniques to Characterize Botulinum Toxin Diffusion
Brief Title: Exploring Advanced Imaging Techniques to Characterize Botulinum Toxin Diffusion in Human Muscle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York Presbyterian Hospital (Other)
Responsible Party: Principal Investigator, Grace Kim, Principal Investigator, Weill Medical College of Cornell University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1002010863
Record Dates: First submitted 2011-08-04; First posted 2011-08-08 (Estimated); Last update posted 2013-10-01 (Estimated); Status verified 2013-09

CONDITIONS: Stroke; Muscle Spasticity
Keywords: MRI; Magnetic Resonance Imaging; Botox; botulinum toxin; neurological; stroke; spasticity; muscle stiffness; diffusion; Weill Cornell; New York Presbyterian Hospital; O'Dell
MeSH Terms: conditions — Stroke; Muscle Spasticity; Neurologic Manifestations | interventions — Botulinum Toxins, Type A; Botulinum Toxins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- botox diffusion (No Intervention): Each subject was given 3 injections in lateral gastrocnemius muscle:2 botox, 1 saline, each injection was 2.5mL. MRI of the lower leg was taken prior to injections and 2 months post for a comparison of diffusion properties.
  Interventions: Drug: Botox (botulinum toxin)

INTERVENTIONS:
Drug: Botox (botulinum toxin) — A series of three injections will be made simultaneously to the gastroc-soleus muscles of the affected lower limb; this will be the only drug intervention/injection session throughout the study, and occurs at baseline. The top injection site, closest to the knee, consists of 25 units of Botox and 0.25 cc saline. The bottom injection site, closest to the ankle, also consists of 25 units of Botox and 0.25 cc saline. The middle injection site will be considered the placebo injection, as it will not contain any Botox (0 units Botox) and 0.25 cc saline.

SUMMARY:
Since the use of botulinum toxin in treating spasticity has already been proven effective, we are now using magnetic resonance imaging to examine the toxin diffusion within muscle (post injection) in order to determine the specific toxin dose required for an optimal treatment response.

DETAILED DESCRIPTION:
Over the past decade, botulinum toxins (BT) have been extensively used to treat any number of diverse disorders, including functionally significant, focal spasticity in the arm and leg of persons with injury/disease of the central nervous system. Spasticity is an involuntary muscle stiffness that limits movement of an extremity and often leads to pain, hygiene problems, difficulty in bed or wheelchair positioning, and functional deficits in self-care and mobility.

There are three BT products on the market: MyoBloc®, Botox®, and Dysport®. FDA approval for use of Botox® in spasticity is anticipated sometime during 2010. In the Weill Cornell Division of Rehabilitation Medicine alone, nearly 50,000 units of Botox® were injected for the treatment of spasticity during the 2008-2009 academic year. (Note: The vast majority of the BT market share in the US rests with Botox®.)

There is excellent evidence supporting the effectiveness of BT in decreasing tone and modest clinical evidence supporting functional improvement. Despite the frequent use, however, there is astonishingly little evidence delineating the impact on diffusion of dosing, dilution, approach to muscle localization, or serotype of BT. To better study these relationships we will be using advanced imaging to develop a model to characterize the physical characteristics of BT diffusion in human skeletal muscle.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of UMN disease
* clinically significant spasticity in the gastrocnemius muscle to warrant Botox® injection (made at the discretion of Dr. O'Dell)
* naïve to all botulinum toxins in the lower extremity

Exclusion Criteria:

* MR incompatibility with implanted ferromagnetic devices.[Specifically, they may not participate in this study if they have a pacemaker, an implanted defibrillator or certain other implanted electronic or metallic devices. They will be screened by the MRI staff for past surgical procedures to determine the possibility of having an implanted medical or metallic device, shrapnel, or other metal, such as metal in the eye.]
* Pregnancy or breast feeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2010-03; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
MRI | Baseline (0 months), 2 months and 3 months
  Subjects will undergo non-contrast MRI's of the target leg prior to Botox injections (0 months), then again at both 2 months and 3 months following the Botox injections.

CONTACTS AND LOCATIONS:
Overall Officials: Michael W O'Dell, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- New York Presbyterian Hospital/Weill Cornell Medical College, New York, New York, United States

REFERENCES:
- See also: NYPH/WCMC Rehabilitation Medicine Research/Trials Site — http://nyp.org/rehab-trials.html